CLINICAL TRIAL: NCT04614428
Title: Tailored, Interventional Health Care Program Designed to Address Seasonal Vulnerability in Patients With Chronic Heart Disease and Multimorbidity: the REsilience to Seasonal ILlness and Increased Emergency admissioNs CarE (RESILIENCE) Trial
Brief Title: Improving Outcomes in Patients With Cardiovascular Seasonality
Acronym: RESILIENCE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sheila Patel (Other Government)
Collaborators: University of Melbourne (Other)
Responsible Party: Sponsor-Investigator, Sheila Patel, Senior Research Fellow, Austin Health
Organization: Austin Health (Other Government)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: CT19026
Record Dates: First submitted 2020-10-29; First posted 2020-11-04 (Actual); Last update posted 2024-03-27 (Actual); Status verified 2024-03

CONDITIONS: Cardiovascular Diseases
MeSH Terms: conditions — Cardiovascular Diseases

STUDY DESIGN:
Intervention Model Description: Randomised control trial of two parallel groups;
  1. Standard Care
  2. Standard Care + RESILIENCE Program
Who Masked: Outcomes Assessor
Masking Description: The people assessing the outcomes will be masked
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard Care Group (No Intervention): Participants will receive the standard care provided by their institution.
- RESILIENCE Program group (Active Comparator): Participants will receive the RESILIENCE Program on top of the standard care provided by their institution.
  Interventions: Behavioral: RESILIENCE Program

INTERVENTIONS:
Behavioral: RESILIENCE Program — In addition to the standard care participants would normally receive (including exposure to any standard hospital avoidance programs), the 150 participants assigned to the RESILIENCE Program group will receive a combination of strategies designed to promote seasonal resilience.
  This includes profiling of seasonal vulnerability; a 60-80 minute home visit by the RESILIENCE Nurse to assess physiological status, behavioural adaptations, environment, and modulating factors; a dedicated RESILIENCE Clinic with a dedicated RESILIENCE physician to develop a long-term plan to help promote/maintain seasonal resilience and; a structured follow-up over the next 12 months to monitor and adjust the participant's status and management from a seasonal perspective.
  Arms: RESILIENCE Program group

SUMMARY:
Despite a range of evidence-based programs to identify high-risk patients and apply strategies to keep them out of hospital, a growing number of cases are "resistant" to such programs. These "seasonal frequent flyers" routinely overwhelm hospital services. The investigators have identified vulnerability to provocation of seasonal and acute weather changes ("seasonality") as a major driver of preventable/costly hospitalisations in typically older patients with heart disease and multimorbidity subject to gold-standard care. From this research the investigators developed the RESILIENCE Program which is tailored to each person and designed to assist the participants to become more "resilient" to changes in the weather.

The overall aim of the RESILIENCE Trial is to demonstrate the cost-effectiveness of an individually tailored, interventional health care program designed to address the debilitating, costly and deadly phenomenon of seasonal vulnerability in a growing number of individuals admitted to hospital with chronic heart disease and multimorbidity.

DETAILED DESCRIPTION:
After informed written consent, a total of 203 participants (of an initially planned 300 participants prior to the COVID pandemic) had comprehensive sociodemographic and clinical profiling to establish extent of multi-morbidity. Baseline demographic, lifestyle and medical history profiling were also completed - including anthropometric measurements, and blood pressure, handgrip strength test and sit-stand tests. The Montreal Cognitive Assessment, depression, anxiety and quality of life questionnaires were also applied. Blood biochemistry will be assessed for vitamin D, blood counts, thyroid and renal function, hemoglobin and glycated hemoglobin levels.

After the initial profiling, 203 participants were randomized to standard care or the RESILIENCE Program group and discharged alive to home.

In addition to the standard care participants would normally receive, the one in two participants assigned to the RESILIENCE Program group will receive a structured follow-up over the next 12 months to monitor and adjust the participant's status and management from a seasonal perspective. These will include a combination of strategies designed to promote seasonal resilience.

Specifically, this will include:

1. Profiling of the participants seasonal vulnerability: prior to hospital discharge, participants will be clinically profiled and then fitted with an physiological monitor (to measure heart rate, physical activity levels) at the point of hospital discharge.
2. Within 7-14 days after discharge a 60-80-minute home visit will be conducted by a dedicated RESILIENCE Nurse to assess:

   * Physiological Status: The physiological monitor will be collected for analysis at this visit and blood pressure will be measured.
   * Environment: A formal home environment assessment including presence/type of heating and/or cooling equipment, air quality and any other factors that might contribute to seasonal instability (e.g. lack of home insulation). Indoor versus outdoor temperature and humidity will also be measured.
   * Behaviour: Participants will be asked to describe the adaptive changes they make to activity levels, diet, clothing and heating/cooling behaviours during winter versus summer and acute weather events; with an immediate assessment relevant to ambient weather conditions.
   * Modulating Factors: The (socio-economic) capacity for the participant/family to apply resources/funds to maintain thermoregulatory control (including clothing choices and ability to pay power bills) throughout the year will be assessed; alongside those personal factors/decisions that potentially determine how they prioritize other forms of expenditure.
3. Participants with the capacity and/or preference for videoconferencing will be offered "virtual/remote" attendance or a standard outpatient clinic appointment at the Austin Hospital RESILIENCE Clinic with a dedicated RESILIENCE physician to develop a long-term plan to help promote/maintain seasonal resilience. The clinic appointments will occur with the individual at 21 days, 6 months and 12 months post hospital discharge.

At 12 months, the comprehensive socio-demographic and clinical profiling will be repeated in the RESILIENCE Program group.

Due to the impact of the COVID epidemic (with extensive lockdowns in Melbourne, Victoria and clinical restrictions at the Austin Hospital), a reduced study cohort was recruited (203 of planned 300 eligible and randomised participants) with follow-up extended beyond 12 months to (partially) restore study power to examine the potential impact of the study intervention on the same health outcomes.

ELIGIBILITY:
Inclusion Criteria:

1. Individual aged 18 years and over.
2. Admitted to hospital due to a medical emergency for any reason but with a chronic form of heart disease (i.e. including. coronary artery disease, atrial fibrillation and/or heart failure) requiring treatment
3. Multimorbidity (defined as two or more chronic conditions requiring active treatment/management).
4. A planned discharge to home within a 10km radius of the hospital.

Exclusion Criteria:

* Living in residential aged care
* Terminal illness and/or unable to give informed consent
* Died during index admission

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 203 (Actual)
Dates: Start 2020-11-25 (Actual); Primary Completion 2023-07-28 (Actual); Study Completion 2023-07-28 (Actual)

PRIMARY OUTCOMES:
Days-alive-out-of-hospital (DAOH) | 12-months (minimum) post randomisation to study census (July 2023)
  Defined as the proportion of maximal days follow-up where the study participant was not admitted to hospital and alive. DAOH data will be collected from hospital records. During minimum 12-month follow-up, the pre-specified threshold for a clinically significant effect in favour of the RESILIENCE Program is a 10% increase in DOAH compared to "standard care".

SECONDARY OUTCOMES:
Overall pattern of hospitalization | 12-months (minimum) post randomisation to study census
  Frequency and causes of unplanned hospitalization plus Emergency Service and out-patient visits and related bed-days will be determined from hospital medical records.
Number of community care visits | 12-months (minimum) post randomisation to study census
  Including visits to the General Practitioner, pharmacist consultations, allied health services, supported-care and pharmacotherapy determined through the RESILIENCE Clinic.
Healthcare costs | 12-months (minimum) post randomisation to study census
  Healthcare costs assessed for extending days-alive-out-of-hospital, transport and other costs due to clinic attendance as well as co-payments for clinic visits and drug therapy.
  All expenditure will be standardized for the reporting year and an extrapolation of the potential impact of the RESILIENCE Program from the perspective of the Australian health care system will be made. QALYs will be calculated from survival and the AQoL-8D as the primary outcome for cost-utility analysis.

CONTACTS AND LOCATIONS:
Overall Officials: Louise M Burrell, MD, Principal Investigator — University of Melbourne
Locations (1):
- Austin Health, Heidelberg, Victoria, Australia

IPD SHARING:
Plan to Share IPD: Yes
Trial data will be disseminated in the form of a publication to a relevant clinical journal and presentation at appropriate scientific conferences. Individual participant data that underlie the published results, may be shared on request by the RESILIENCE TRIAL Investigators at the completion of the trial and reporting of the endpoints.
Supporting Information: Study Protocol
Time Frame: Beginning following main results publication; no end date determined
Access Criteria: Case-by-case basis at the discretion of the Primary Sponsor and RESILIENCE TRIAL Investigators and provide a methodologically sound proposal.

REFERENCES:
- [Derived] Stewart S, Patel SK, Lancefield TF, Sampaio Rodrigues T, Doumtsis N, Moini N, Harley A, Vaughan-Fowler ER, Chan YK, Chen A, Chye D, Liew DF, McMaster C, Ramchand J, Yates PA, Kwong JC, McDonald CF, Burrell LM. Promoting resilience to weather-related and seasonal provocations to health in people with multimorbid heart disease: a prospective pragmatic, randomised trial. Med J Aust. 2025 Jul 21;223(2):77-84. doi: 10.5694/mja2.52699. Epub 2025 Jun 24. PMID 40556316
- [Derived] Stewart S, Patel SK, Lancefield TF, Rodrigues TS, Doumtsis N, Jess A, Vaughan-Fowler ER, Chan YK, Ramchand J, Yates PA, Kwong JC, McDonald CF, Burrell LM. Vulnerability to environmental and climatic health provocations among women and men hospitalized with chronic heart disease: insights from the RESILIENCE TRIAL cohort. Eur J Cardiovasc Nurs. 2024 Apr 12;23(3):278-286. doi: 10.1093/eurjcn/zvad076. PMID 37625011